CLINICAL TRIAL: NCT06572267
Title: Safety and Efficacy of Meplazumab in Patients With Coronary Artery Disease: a Single-center, Placebo-controlled, Exploratory, Phase 2, Pilot Trial
Brief Title: Safety and Efficacy of Meplazumab in Patients With Coronary Artery Disease
Acronym: REC-SAFECAD
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Xijing Hospital (Other)
Responsible Party: Principal Investigator, Ling Tao, MD, PhD, Director of the Department of Cardiology, Xijing Hospital
Allocation: Randomized | Model: Sequential | Masking: Single | Purpose: Treatment
Other Study IDs: KY20242170-F-1
Record Dates: First submitted 2024-08-22; First posted 2024-08-27 (Actual); Last update posted 2026-01-23 (Actual); Status verified 2026-01

CONDITIONS: Coronary Artery Disease
Keywords: Meplazumab; coronary artery disease; inflammation; lipid deposition
MeSH Terms: conditions — Coronary Artery Disease; Inflammation | interventions — mepolizumab; Population Groups; Sodium Chloride

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Mepolizumab low dose group (Experimental): Mepolizumab (Jiangsu Pacific Menok Biopharmaceutical Co), 0.05 mg/kg, monthly.
  Meperizumab was dissolved in 1 mL of sterile water and added to 100 mL of saline for intravenous infusion. The intravenous infusion shall be completed within 30 to 60 min.
  Interventions: Drug: Mepolizumab low dose group
- Mepolizumab middle dose group (Experimental): Mepolizumab (Jiangsu Pacific Menok Biopharmaceutical Co), 0.1 mg/kg, monthly.
  Meperizumab was dissolved in 1 mL of sterile water and added to 100 mL of saline for intravenous infusion. The intravenous infusion shall be completed within 30 to 60 min.
  Interventions: Drug: Mepolizumab middle dose group
- Mepolizumab high dose group (Experimental): Mepolizumab (Jiangsu Pacific Menok Biopharmaceutical Co), 0.2 mg/kg, monthly.
  Meperizumab was dissolved in 1 mL of sterile water and added to 100 mL of saline for intravenous infusion. The intravenous infusion shall be completed within 30 to 60 min.
  Interventions: Drug: Mepolizumab high dose group
- Placebo group (Placebo Comparator): Saline, 100 ml, intravenous infusion
  Interventions: Drug: Saline

INTERVENTIONS:
Drug: Mepolizumab low dose group — Meperizumab (0.05 mg/kg) was dissolved in 1 mL of sterile water and added to 100 mL of saline for intravenous infusion. The intravenous infusion shall be completed within 30 to 60 min.
  Arms: Mepolizumab low dose group
Drug: Mepolizumab middle dose group — Meperizumab (0.1 mg/kg) was dissolved in 1 mL of sterile water and added to 100 mL of saline for intravenous infusion. The intravenous infusion shall be completed within 30 to 60 min.
  Arms: Mepolizumab middle dose group
Drug: Mepolizumab high dose group — Meperizumab (0.2 mg/kg) was dissolved in 1 mL of sterile water and added to 100 mL of saline for intravenous infusion. The intravenous infusion shall be completed within 30 to 60 min.
  Arms: Mepolizumab high dose group
Drug: Saline — Intravenous infusion of saline 100 mL shall be completed within 30 to 60 min.
  Arms: Placebo group

SUMMARY:
The development of coronary atherosclerosis is closely related to inflammation, and CD147 may play an important role in its process. The present study was designed to evaluate the effects of long-term administration of mepolizumab (humanized anti-CD147 antibody) on lipid deposition and inflammation in coronary atherosclerotic plaques in patients with high-risk coronary artery disease, and to preliminarily explore the efficacy, safety, and dosage of long-term administration of mepolizumab in this population.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with chronic coronary syndrome
2. Non-target lesions with stenosis ≥50% by visual assessment
3. Angina symptoms manageable via antianginal medication
4. High attenuation coefficient (≥-70.1 HU) of perivascular adipose tissue (PVAT) around non-target lesions as assessed by coronary CT angiography (CCTA)
5. Patients who are able to complete the follow-up and compliant to the prescribed medication

Exclusion Criteria:

1. Under the age of 18
2. Unable to give informed consent or currently participating in another trial and not yet at its primary endpoint
3. Patient is a woman who is pregnant or nursing (a pregnancy test must be performed within 7 days prior to the index procedure in women of child-bearing potential according to local practice)
4. Concurrent medical condition with a life expectancy of less than 3 years
5. Haemodynamical unstable
6. Known contraindications to medications such as test drug and its components, heparin, or contrast
7. The following criteria are met for any of the laboratory test indicators at the time of screening ①ALT/AST >3ULN；②TBil ≥2ULN；③WBC>2ULN；④NEUT<0.5×109 /L；⑤PLT<30×109 /L；⑥eGFR <60 mL/min/1.73 m2（CKD-EPI formula）
8. Suffering from severe systemic diseases, tumors, immune system disorders, infections, malignancy, which in the opinion of the investigator make participation in this study inappropriate

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18 (Estimated)
Dates: Start 2024-10-16 (Actual); Primary Completion 2026-09-01 (Estimated); Study Completion 2027-03-01 (Estimated)

PRIMARY OUTCOMES:
Proportion of high PVAT attenuation coefficient among non-target lesion(s) | 6 months
  Proportion of high PVAT attenuation coefficient (≥-70.1 HU) among non-target lesion(s) assessed by CCTA

SECONDARY OUTCOMES:
Change in PVAT attenuation coefficient of non-target lesion(s) from baseline to follow-up | 6 months
Change in non-target lesion plaque composition as assessed by CCTA from baseline to follow-up | 6 months
Changes in inflammatory biomarkers from baseline to follow-up | 6 months
  Biomarkers including hs-CRP, IL-1, IL-2, IL-4, IL-6, INF-α, IL-8, IL-10, IL-12p70, IL-17, IL-1β, TNF-α and IFN-γ
Device-oriented clinical endpoint (DoCE) | 1 month and 6 months
  Device-oriented clinical endpoint is a composite endpoint including cardiac death, target vessel infarction, and clinically driven target lesion revascularization
Cardiac death | 1 month and 6 months
  The individual component of the DoCE
Target vessel infarction | 1 month and 6 months
  The individual component of the DoCE
Clinically driven target lesion revascularization | 1 month and 6 months
  The individual component of the DoCE
Patient-oriented composite endpoint (PoCE) | 1 month and 6 months
  Patient-oriented composite endpoint is a composite endpoint including all-cause death, any stroke, any myocardial infarctions, and any revascularization
All-cause death | 1 month and 6 months
  The individual component of the PoCE
Any stroke | 1 month and 6 months
  The individual component of the PoCE
Any myocardial infarction | 1 month and 6 months
  The individual component of the PoCE
Any revascularization | 1 month and 6 months
  The individual component of the PoCE
Changes in gene expression of peripheral blood mononuclear cells | 6 months
Any adverse events | 1, 2, 3, 4, 5, and 6 months
  All adverse events (AE) will be recorded and categorized according to CTCAE Ver 5.0

CONTACTS AND LOCATIONS:
Overall Officials: Ling Tao, M.D., Ph.D., Study Chair — Xijing Hospital; Ping Zhu, M.D., Ph.D., Study Chair — Xijing Hospital; Chao Gao, M.D., Ph.D., Study Chair — Xijing Hospital
Locations (1):
- Ling Tao, Xi'an, Shannxi, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Sturhan H, Ungern-Sternberg SN, Langer H, Gawaz M, Geisler T, May AE, Seizer P. Regulation of EMMPRIN (CD147) on monocyte subsets in patients with symptomatic coronary artery disease. Thromb Res. 2015 Jun;135(6):1160-4. doi: 10.1016/j.thromres.2015.03.022. Epub 2015 Mar 20. PMID 25824988
- [Background] Lv JJ, Wang H, Zhang C, Zhang TJ, Wei HL, Liu ZK, Ma YH, Yang Z, He Q, Wang LJ, Duan LL, Chen ZN, Bian H. CD147 Sparks Atherosclerosis by Driving M1 Phenotype and Impairing Efferocytosis. Circ Res. 2024 Jan 19;134(2):165-185. doi: 10.1161/CIRCRESAHA.123.323223. Epub 2024 Jan 3. PMID 38166463